CLINICAL TRIAL: NCT06167122
Title: Long-term Follow-up and Treatment Protocol for Craniofacial Fibrous Dysplasia From 40-year Data at Chang Gung Memorial Hospital: A Retrospective Case Series
Brief Title: Treatment Protocol and Long-Term Outcomes in Craniofacial Fibrous Dysplasia
Acronym: CFD
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Pangyunchou, Associate Professor, Chang Gung Memorial Hospital
Other Study IDs: 202000158B0
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Craniofacial Fibrous Dysplasia
Keywords: Craniofacial fibrous dysplasia; Optic nerve decompression; Hormone therapy
MeSH Terms: conditions — Craniofacial Fibrous Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Craniofacial fibrous dysplasia: Fibro-osseous lesions within the affected bones based on image, and surgical intervention based on 4 different anatomical zones.
  Interventions: Procedure: Craniofacial reconstruction

INTERVENTIONS:
Procedure: Craniofacial reconstruction — Zone 1 lesions: radical excision and immediate reconstruction with bone grafts for fibrous dysplasia lesions.
  Zone 2 lesions: trimming & recontouring. Zone 3 lesions: observation or conservative recontouring; optic nerve decompression performed when continuous deterioration of vision, and external auditory canal surgery performed when cholesteatoma/near total ear canal stenosis.
  Zone 4: observation or conservative recontouring; orthognathic surgery performed when malocclusion or midface retrusion noted.

SUMMARY:
Craniofacial fibrous dysplasia (CFD) is a nonneoplastic disease characterized by fibro-osseous lesions in the affected bones. Treatment is mainly surgical and is stratified based on four different anatomical zones. This study aimed to evaluate the long-term outcomes and refine the algorithm for CFD.

DETAILED DESCRIPTION:
According to Chen et. al for the appropriate surgical management of FD the craniofacial skeleton can be divided into four zones according to the consideration of facial cosmesis, vital anatomical region and function preserving. The aim of the study was to evaluate the outcome of nearly 40 years long-term follow up cohort group and refine the algorithm of surgical intervention of FD under 4 zones classification.

ELIGIBILITY:
Inclusion Criteria:

* Received CFD surgical intervention between 1972 and 2019
* Personal interviews: between late 2019 and 2020, covering a postoperative period of over 20 years
* All the surgery were performed by a senior surgeon (Yu-Ray Chen) at Chang Gung Craniofacial Center

Exclusion Criteria:

* Patients who underwent surgical treatment at other institutions during the follow-up period or those who did not return to the craniofacial outpatient department for follow-up and receive computed tomography scans between 2019 and 2020 will be excluded.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patient with craniofacial fibrous dysplasia, and received craniofacial surgery
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-03-14 (Actual)

PRIMARY OUTCOMES:
Recurrence | Personal interviews with facial bone computed tomography obtained on late 2019 and 2020
  Recurrence based on facial bone computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Pang-Yun Chou, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No